CLINICAL TRIAL: NCT05241470
Title: A Phase 2 Multi-Center, Randomized, Double Masked, Placebo Controlled Study to Assess the Safety and Efficacy of ST-100 Ophthalmic Solution in Subjects Diagnosed With Dry Eye Disease
Brief Title: Study of ST-100 as Treatment for Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stuart Therapeutics, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST100-001
Record Dates: First submitted 2022-01-05; First posted 2022-02-15 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose ST-100 Ophthalmic Solution (Active Comparator): Low Dose ST100-001 Ophthalmic solution, 20mcg/ml
  Interventions: Drug: ST-100 Ophthalmic Solution
- High Dose ST-100 Ophthalmic Solution (Active Comparator): High Dose ST100-001 Ophthalmic Solution, 50mcg/ml
  Interventions: Drug: ST-100 Ophthalmic Solution
- Placebo Ophthalmic Solution (Placebo Comparator): Placebo Ophthalmic Solution (vehicle)
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: ST-100 Ophthalmic Solution — One drop in each eye twice a day
  Other Names: ST-100
  Arms: High Dose ST-100 Ophthalmic Solution; Low Dose ST-100 Ophthalmic Solution
Drug: Placebo Ophthalmic Solution — One drop in each eye twice a day
  Other Names: Vehicle
  Arms: Placebo Ophthalmic Solution

SUMMARY:
The objective of this study is to compare the safety and efficacy of two different concentrations of ST-100 Ophthalmic Solution to placebo (vehicle) for the treatment of the signs and symptoms of dry eye.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, double-masked, randomized, placebo-controlled clinical study. Subjects will be randomized to one of the following treatment arms at Visit 2 (Day 1):

* Low dose ST-100 Ophthalmic Solution: 1 drop twice daily (BID) in each eye
* High dose ST-100 Ophthalmic Solution: 1 drop BID in each eye
* Placebo Ophthalmic Solution (Vehicle): 1 drop BID in each eye

Approximately 150 subjects will be randomly assigned to one of the three groups (1:1:1) to receive either ST-100 Ophthalmic Solution or placebo solution as topical ophthalmic drops administered bilaterally BID for 4 weeks. Subjects, Sponsor, Contract Research Organization (CRO), and site personnel will be masked to treatment assignment.

The clinical hypotheses for this study is that low dose and high dose ST-100 Ophthalmic Solution twice daily (BID) is superior to its vehicle (BID) for the primary endpoints of signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a subject reported history of dry eye;
* Have a history of use of eye drops for dry eye symptoms;
* Have symptoms of dry eye as determined by Ocular Discomfort & 4-symptom questionnaire;
* Have a Schirmer's Test score of ≤ 10 mm and ≥ 1 mm;
* Have conjunctival redness;
* Have corneal fluorescein staining;
* Have lissamine green conjunctival staining;
* Have signs and symptoms responses to Controlled Adverse Environment (CAE®);

Exclusion Criteria:

* Have any clinically significant slit lamp findings;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation ;
* Have worn contact lenses;
* Have used any eye drops;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery
* Have used Restasis, Xiidra, or Cequa ophthalmic solutions
* Have any planned ocular and/or lid surgeries or any ocular surgery;
* Have used, are using or anticipate using permanent or temporary punctal plugs during the study;
* Be currently taking any topical ophthalmic prescription;
* Be currently taking or have taken Omega-3 supplements;
* Be unable to read an eye chart;
* Be a woman who is pregnant, nursing, or planning a pregnancy;
* Be unwilling to submit a urine pregnancy test (or early termination visit) if of childbearing potential;
* Be a woman of childbearing potential who is not using an acceptable means of birth control;
* Have a known allergy and/or sensitivity to the test article or its components;
* Have a condition or be in a situation that the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device;
* Be currently using any medication known to cause ocular drying that is not used on a stable dosing regimen;
* Have a known history of meibomian gland procedures (e.g., LipiFlow, LPI, probing, etc.);
* Be unable or unwilling to follow instructions, including participation in all study assessments and visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Baratta, MD, Study Chair — Stuart Therapeutics, Inc.
Locations (3):
- United States (3):
  - Andover Eye Associates, Andover, Massachusetts
  - Andover Eye Associates - Raynham, Raynham, Massachusetts
  - Total Eye Care, P.A., Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants participated in the run-in phase of the study before randomization.
Units Other Than Participants: Eyes
Groups:
- Run-In: Run-In Phase
Period: Placebo Run-In
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution | Run-In
Started | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 160; 320 Eyes
Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 160; 320 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes
Period: Randomized Study
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution | Run-In
Started | 53; 106 Eyes | 53; 106 Eyes | 54; 108 Eyes | 0; 0 Eyes
Completed | 48; 96 Eyes | 50; 100 Eyes | 48; 96 Eyes | 0; 0 Eyes
Not Completed | 5; 10 Eyes | 3; 6 Eyes | 6; 12 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Low Dose ST-100 Ophthalmic Solution: Low Dose ST100-001 Ophthalmic solution, 20mg/ml
  ST-100 Ophthalmic Solution: One drop in each eye twice a day
- High Dose ST-100 Ophthalmic Solution: High Dose ST100-001 Ophthalmic Solution, 50mg/ml
  ST-100 Ophthalmic Solution: One drop in each eye twice a day
- Total: Total of all reporting groups
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution | Total
Number analyzed (Participants) | 53 | 53 | 54 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.29) | 61.9 (11.60) | 63.4 (13.28) | 63.2 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 29 | 43 | 112
  Male | 13 | 24 | 11 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 15 | 15 | 18 | 48
  White | 35 | 38 | 36 | 109
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Total Corneal Fluorescein Staining [Mean (Standard Deviation); unit: units on a scale] — The fluorescein staining is graded with the Ora Calibra® Corneal and Conjunctival Staining Scale. The scale is used to evaluate inferior, superior, central, temporal, and nasal region. Staining in each region is graded 0 to 4 where 0 means no staining, and 4 means worst staining. Higher score indicates more staining. The corneal sum score is the sum from the inferior, superior, and central regions (min 0, max 12). The conjunctival sum score is the sum of scores from the nasal and temporal regions (min 0, max 8). The total eye score is the sum of scores from all five regions (min 0, max 20).
  units on a scale | 4.78 (0.781) | 4.86 (1.094) | 4.81 (0.928) | 4.82 (0.937)
Ocular Discomfort Scale [Mean (Standard Deviation); unit: units on a scale] — Ocular Discomfort Scale is graded using the Ora Calibra Ocular Discomfort Scale (ODS). The scale ranges from 0 means no discomfort to 4 means worst discomfort. Higher score indicates more discomfort.
  units on a scale | 2.6 (1.06) | 2.4 (1.04) | 2.5 (1.11) | 2.5 (1.07)
Unanesthetized Schirmer's test [Mean (Standard Deviation); unit: mm] | 4.4 (2.77) | 5.2 (2.84) | 5.0 (2.87) | 4.9 (2.83)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Total Corneal Fluorescein Staining (Ora Calibra® Scale) in the Study Eye at Visit 7 (Day 29) Pre-Controlled Adverse Environment (Pre-CAE)
Description: The fluorescein staining is graded with the Ora Calibra® Corneal and Conjunctival Staining Scale. The scale is used to evaluate 3 corneal regions. Staining in each region is graded 0 to 4 where 0 means no staining, and 4 means worst staining. Higher score indicates more staining. The scoring reported ranges from 0-12. Mean change from baseline was calculated.
Time Frame: Visit 2 (Day 1) to Visit 7 (Day 29)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: Study Eye
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 53 | 53 | 54
Number analyzed (Study Eye) | 53 | 53 | 54
units on a scale | -0.17 (0.186) | -0.17 (0.182) | -0.18 (0.185)
Statistical Analysis 1: Comparison: Low Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.9575, ANCOVA; Mean Difference (Net) = 0.01
Statistical Analysis 2: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.9741, ANCOVA; Mean Difference (Net) = 0.01

2. Primary Outcome: Change From Baseline of Ocular Discomfort in the Study Eye at Visit 7 (Day 29) Pre-CAE
Description: Ocular Discomfort Scale is graded using the Ora Calibra Ocular Discomfort Scale (ODS). The scale ranges from 0 means no discomfort to 4 means worst discomfort. Higher score indicates more discomfort.
Time Frame: Visit 2 (Day 1) to Visit 7 (Day 29)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Study Eye
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 53 | 53 | 54
Number analyzed (Study Eye) | 53 | 53 | 54
score on a scale | -0.3 (0.14) | -0.4 (0.13) | -0.3 (0.14)
Statistical Analysis 1: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.5696, ANCOVA

3. Secondary Outcome: Unanesthetized Schirmer's Responder Rate
Description: The Schirmer's test strip is placed in the lower temporal lid margin of each eye. After 5 minutes, the test strip is removed and the length of the moistened area will be recorded in millimeters (mm) for each eye. The percentage of responders who had ≥ 10 mm increase from baseline in study eye in unanesthetized Schirmer's test was recorded.
Time Frame: Visit 7 (Day 29), Pre-CAE
Population: The measurements are reported for each visit. The number of subjects in each group varied at each visit. The overall analyzed number of participants are from the ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 53 | 53 | 54
Participants | 48 | 49 | 48
Statistical Analysis 1: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.0266, Fisher Exact

4. Secondary Outcome: Change From Baseline of Best-Corrected Visual Acuity (ETDRS) - logMAR (Fellow Eye) at Visit 3 (Day 2)
Description: LogMAR visual acuity (VA) is assessed using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The last line in which a letter is read correctly will be taken as the base logMAR reading. To this value will be added the number "N x 0.02" where 'N' represents the total number of letters missed up to and included in the last line read. This total sum represents the logMAR VA for that eye.
Time Frame: Visit 3 (Day 2)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Fellow Eye
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 52 | 53 | 54
Number analyzed (Fellow Eye) | 52 | 53 | 54
logMAR | -0.003 (0.0104) | -0.028 (0.0104) | 0013 (0.0103)
Statistical Analysis 1: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.0055, ANCOVA

5. Secondary Outcome: Change From Baseline to Visit 4 (Day 4) in Ocular Surface Disease Index (Blurred Vision)
Description: Ocular Surface Disease Index (OSDI) Questions 4: Have you experienced blurred vision during the last week? on 0-4 Scale where 4 is the worst at pre-CAE®
Time Frame: Visit 4 (Day 4), Non-CAE
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Study Eye
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 53 | 53 | 54
Number analyzed (Study Eye) | 53 | 53 | 54
score on a scale | -0.1 (0.12) | -0.3 (0.12) | 0.2 (0.12)
Statistical Analysis 1: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.0097, ANCOVA

6. Secondary Outcome: Change From Baseline to Visit 6 (Day 15) in Ocular Surface Disease Index (Pain)
Description: Ocular Surface Disease Index (OSDI) Questions 3: Have you experienced painful or sore eyes during the last week? on 0-4 Scale where 4 is the worst at pre-CAE®
Time Frame: Visit 6 (Day 15) Pre-CAE
Population: The measurements are reported for each visit. The number of subjects in each group varied slightly at each visit. The overall number analyzed are reported based on the ITT population.
  -
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Study Eye
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 49 | 51 | 49
Number analyzed (Study Eye) | 49 | 51 | 49
score on a scale | -0.1 (0.11) | -0.4 (0.11) | 0.0 (0.11)
Statistical Analysis 1: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.0137, ANCOVA

7. Secondary Outcome: Change From Baseline in Ocular Discomfort Assessed by 4-Symptom Questionnaire
Description: The Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire is used, which includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging. Each symptom rating ranges from 0 to 5, where 0 = None and 5 = Worst. Higher score means worse symptom. Min score = 0, max score = 25.
Time Frame: Visit 6 (Day 15) Pre-CAE
Population: The measurements are reported for each visit. The number of subjects in each group varied slightly at each visit. The overall analyzed number of participants were from the ITT population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Study Eye
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 49 | 51 | 49
Number analyzed (Study Eye) | 49 | 51 | 49
score on a scale | -0.2 (0.11) | -0.4 (0.11) | 0.0 (0.11)
Statistical Analysis 1: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.0332, ANCOVA

8. Post Hoc Outcome: Change From Baseline in Fluorescein Staining in the Total Eye Sum - Both Eyes Together
Description: The fluorescein staining is graded with the Ora Calibra® Corneal and Conjunctival Staining Scale. The scale is used to evaluate inferior, superior, central, temporal, and nasal region. Staining in each region is graded 0 to 4 where 0 means no staining, and 4 means worst staining. Higher score indicates more staining. The corneal sum score is the sum of scores from the inferior, superior, and central regions (min 0, max 12). The conjunctival sum score is the sum of scores from the nasal and temporal regions (min 0, max 8). The total eye score is the sum of scores from all five regions (min 0, max 20). The average values of both eyes assessment were reported (min 0, max 20)
Time Frame: Visit 7 (Day 28) Pre CAE
Population: The analysis was done on both study and fellow eyes combined
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 50 | 48 | 48
Number analyzed (Eyes) | 100 | 96 | 96
units on a scale | -0.33 (1.660) | -0.42 (1.810) | 0.16 (2.075)
Statistical Analysis 1: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.0394, t-test, 2 sided

9. Post Hoc Outcome: Change From Baseline in Fluorescein Staining in Conjunctival Sum - Both Eyes Together
Description: as for outcome 8
Time Frame: Visit 7 (Day 28), Pre CAE
Population: The analysis was done on both study and fellow eyes combined
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Total Eyes
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 50 | 48 | 48
Number analyzed (Total Eyes) | 100 | 96 | 96
units on a scale | -0.01 (0.793) | -0.14 (1.057) | 0.17 (1.007)
Statistical Analysis 1: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.0121, Wilcoxon (Mann-Whitney)

10. Post Hoc Outcome: Change From Baseline in Fluorescein Staining in the Temporal Region - Both Eyes Together
Description: The fluorescein staining is graded with the Ora Calibra® Corneal and Conjunctival Staining Scale. The scale is used to evaluate inferior, superior, central, temporal, and nasal region. Staining in each region is graded 0 to 4 where 0 means no staining, and 4 means worst staining. Higher score indicates more staining. This assessment reported the staining score in temporal region using the Corneal and Conjunctival Fluorescein Staining Scale (min 0, max 4). The average values of both eyes assessment were reported (min 0, max 4).
Time Frame: Visit 7 (Day 28), Pre-CAE
Population: The count is based on the study and fellow eyes combined
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Total Eyes
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 50 | 48 | 48
Number analyzed (Total Eyes) | 100 | 96 | 96
units on a scale | -0.07 (0.479) | -0.07 (0.644) | 0.12 (0.593)
Statistical Analysis 1: Comparison: High Dose ST-100 Ophthalmic Solution vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.0224, Wilcoxon (Mann-Whitney)

11. Post Hoc Outcome: Change From Baseline in Ocular Discomfort Scale (Ora Calibra Scale) During the CAE - Area Under the Curve
Description: Ocular Discomfort Scale is graded using the Ora Calibra Ocular Discomfort Scale (ODS). The scale ranges from 0 means no discomfort to 4 means worst discomfort. Higher score indicates more discomfort. Area under the curve is presented. AUC at each visit is calculated as follows: Calculate (time point - previous time point)*0.5*(discomfort score at time point + previous discomfort score at time point) then sum all of those values together. Given that this was taken every 5 minutes from 0 to 90 minutes, the maximum value for AUC would then be (5*0.5*8)*18=360, and the minimum value would be (5*0.5*0)*18=0. Given this, the minimum and maximum change from baseline would be -360 to 360.
Time Frame: Baseline, Visit 5 (Day 7), Visit 6 (Day 14), and Visit 7 (Day 28)
Population: Analysis was done on ITT population with Observed Data Only. The number analyzed in one or more rows differs from overall number analyzed because the number of participants/study eye analyzed can vary with each visit.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale*min
Units Other Than Participants: Study Eye
Groups:
- Low Dose ST-100 Ophthalmic Solution: Low Dose ST100-001 Ophthalmic solution, 20mcg/ml ST-100 Ophthalmic Solution: One drop in each eye twice a day
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 53 | 53 | 54
Number analyzed (Study Eye) | 53 | 53 | 54
Score on a scale*min
  Change from Baseline to Visit 5 (Day 7), 5 Minutes: number analyzed (Participants) | 49 | 53 | 54
  Change from Baseline to Visit 5 (Day 7), 5 Minutes: number analyzed (Study Eye) | 49 | 53 | 54
  Change from Baseline to Visit 5 (Day 7), 5 Minutes | -0.76 (0.511) | -1.05 (0.501) | -0.18 (0.506)
  Change from Baseline to Visit 5 (Day 7), 45 Minutes: number analyzed (Participants) | 49 | 53 | 54
  Change from Baseline to Visit 5 (Day 7), 45 Minutes: number analyzed (Study Eye) | 49 | 53 | 54
  Change from Baseline to Visit 5 (Day 7), 45 Minutes | -6.98 (3.791) | -13.10 (3.713) | -5.39 (3.743)
  Change from Baseline to Visit 5 (Day 7), 90 Minutes: number analyzed (Participants) | 49 | 53 | 54
  Change from Baseline to Visit 5 (Day 7), 90 Minutes: number analyzed (Study Eye) | 49 | 53 | 54
  Change from Baseline to Visit 5 (Day 7), 90 Minutes | -9.82 (6.570) | -17.43 (6.430) | -5.70 (6.487)
  Change from Baseline to Visit 6 (Day 14), 5 Minutes: number analyzed (Participants) | 48 | 48 | 49
  Change from Baseline to Visit 6 (Day 14), 5 Minutes: number analyzed (Study Eye) | 48 | 48 | 49
  Change from Baseline to Visit 6 (Day 14), 5 Minutes | 0.13 (0.542) | -1.54 (0.542) | -0.30 (0.537)
  Change from Baseline to Visit 6 (Day 14), 45 Minutes: number analyzed (Participants) | 48 | 48 | 49
  Change from Baseline to Visit 6 (Day 14), 45 Minutes: number analyzed (Study Eye) | 48 | 48 | 49
  Change from Baseline to Visit 6 (Day 14), 45 Minutes | -8.15 (3.727) | -16.46 (3.729) | -9.36 (3.683)
  Change from Baseline to Visit 6 (Day 14), 90 Minutes: number analyzed (Participants) | 48 | 48 | 49
  Change from Baseline to Visit 6 (Day 14), 90 Minutes: number analyzed (Study Eye) | 48 | 48 | 49
  Change from Baseline to Visit 6 (Day 14), 90 Minutes | -9.32 (6.621) | -22.34 (6.619) | -16.89 (6.539)
  Change from Baseline to Visit 7 (Day 28), 5 Minutes: number analyzed (Participants) | 48 | 50 | 48
  Change from Baseline to Visit 7 (Day 28), 5 Minutes: number analyzed (Study Eye) | 48 | 50 | 48
  Change from Baseline to Visit 7 (Day 28), 5 Minutes | -0.28 (0.576) | -1.49 (0.565) | -0.77 (0.576)
  Change from Baseline to Visit 7 (Day 28), 45 Minutes: number analyzed (Participants) | 48 | 50 | 48
  Change from Baseline to Visit 7 (Day 28), 45 Minutes: number analyzed (Study Eye) | 48 | 50 | 48
  Change from Baseline to Visit 7 (Day 28), 45 Minutes | -8.58 (4.676) | -19.27 (4.578) | -11.18 (4.661)
  Change from Baseline to Visit 7 (Day 28), 90 Minutes: number analyzed (Participants) | 48 | 50 | 48
  Change from Baseline to Visit 7 (Day 28), 90 Minutes: number analyzed (Study Eye) | 48 | 50 | 48
  Change from Baseline to Visit 7 (Day 28), 90 Minutes | -17.64 (8.266) | -32.20 (8.085) | -21.48 (8.238)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 month
Description: Safety population: 52 in low dose, 53 in high dose, 54 in Placebo. ST-100 was safe and well tolerated in the study. There were no meaningful imbalances among treatment groups in either ocular or non-ocular treatment emergent adverse events. All serious adverse events were considered unexpected and not related to study drug. Other AEs > 5% (reduced VA and instillation site pain) were seen in one or at most two early visits but were no longer seen in the same patients as the trial progressed.
Arm/Group | Low Dose ST-100 Ophthalmic Solution | High Dose ST-100 Ophthalmic Solution | Placebo Ophthalmic Solution | Run-In
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53 | 1/54 | 0/160
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/53 | 2/54 | 0/160
Other Adverse Events (participants affected / at risk) | 6/52 | 6/53 | 8/54 | 0/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose ST-100 Ophthalmic Solution (N=52) | High Dose ST-100 Ophthalmic Solution (N=53) | Placebo Ophthalmic Solution (N=54) | Run-In (N=160)
Respiratory Depression related to congestive heart failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Poor organ function (General disorders) | 0 | 0 | 1 | 0 — Kidney, heart, liver
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose ST-100 Ophthalmic Solution (N=52) | High Dose ST-100 Ophthalmic Solution (N=53) | Placebo Ophthalmic Solution (N=54) | Run-In (N=160)
Visual acuity reduced (Eye disorders) | 2 | 3 | 3 | 0
Instillation site pain (General disorders) | 4 | 3 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05241470/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT05241470/SAP_001.pdf